CLINICAL TRIAL: NCT04971733
Title: An Open-Label Phase 1b/2 Study to Assess Safety and Target Engagement of E2814 in Subjects With Mild to Moderate Cognitive Impairment Due to Dominantly Inherited Alzheimer's Disease
Brief Title: A Study to Assess Safety and Target Engagement of E2814 in Participants With Mild to Moderate Cognitive Impairment Due to Dominantly Inherited Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: E2814-G000-103; 2020-005728-12 (EudraCT Number)
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: E2814; Alzheimer disease; Dominantly inherited Alzheimer disease; Mild and moderate cognitive impairment; Central nervous system disease
MeSH Terms: conditions — Alzheimer Disease; Lymphoma, Follicular; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A, Phase 1b and 2: E2814 (Experimental): Participants will receive E2814 as an intravenous infusion at set intervals over 12 weeks in Phase 1b and over 96 weeks in Phase 2.
  Interventions: Drug: E2814
- Cohort B: E2814 (Experimental): Participants will receive E2814 as an intravenous infusion at set intervals over 52 weeks.
  Interventions: Drug: E2814

INTERVENTIONS:
Drug: E2814 — E2814 intravenous infusion.

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of intravenous (IV) infusions of E2814 in participants with dominantly inherited Alzheimer's disease (DIAD), and to evaluate target engagement (TE) of E2814 on microtubule binding region (MTBR)-tau species in cerebrospinal fluid (CSF) in participants with DIAD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 80 years at the time of informed consent
2. Individuals who are confirmed to be mutation positive for presenilin 1 (PSEN1), amyloid precursor protein (APP), or presenilin 2 (PSEN2) gene that is associated with DIAD
3. Clinical Dementia Rating - Sum of Boxes (CDR-SB) score 5 to 12 at Screening
4. Able to undergo magnetic resonance imaging (MRI), lumbar puncture (LP), PET, and complete all study-related testing and evaluations
5. Has a study partner who in the investigator's judgment is able to provide accurate information as to the participant's cognitive and functional abilities, who agrees to provide information at the study visits which require informant input for scale completion

Exclusion Criteria:

1. Clinically significant illness that required medical treatment within 8 weeks before the 1st dose or a clinically significant infection that required medical treatment within 4 weeks before 1st dose
2. Females who are breastfeeding or pregnant at Screening or Baseline
3. Females of childbearing potential who:

   Within 3 months before screening, did not use a highly effective method of contraception
4. Any neurological condition that may be contributing to cognitive impairment above and beyond that caused by the participant's Alzheimer's disease (AD)
5. History of transient ischemic attacks, stroke, or seizures within 12 months of Screening
6. History of clinically important carotid or vertebrobasilar stenosis, plaque, or other prominent risk factor for stroke or cerebral haemorrhage (including atrial fibrillation and anticoagulation). Low dose aspirin (less than or equal to [<=] 325 milligram [mg] daily) is not exclusionary
7. Any current psychiatric diagnosis or symptoms, (example, hallucinations, major depression, or delusions) that could interfere with study procedures in the participant
8. Geriatric Depression Scale (GDS) score greater than or equal to 8 at Screening
9. Contraindications to MRI scanning, including but not limited to pacemaker/cardiac defibrillator, neurostimulators, ferromagnetic metal implants (example, in skull and cardiac devices other than those approved as safe for use in MRI scanners)
10. Evidence of other clinically significant lesions on brain MRI at Screening that could indicate a dementia diagnosis other than AD
11. Other significant pathological findings on brain MRI at Screening
12. Hypersensitivity to E2814 or any of the excipients, or to any monoclonal antibody (mAb) treatment
13. Any immunological disease which is not adequately controlled, or which requires treatment with immunoglobulins, systemic monoclonal antibodies (or derivatives of monoclonal antibodies), systemic immunosuppressants, or plasmapheresis during the study
14. With a bleeding disorder of current chronic use of anticoagulants (example, warfarin, dabigatran, rivaroxaban or apixaban) or of clopidogrel is exclusionary. Limited (occasional or isolated) use of anticoagulants/antiplatelet compounds in cases such as surgical procedures
15. Have thyroid stimulating hormone outside of normal range. Other tests of thyroid function with results outside the normal range should only be exclusionary if they are considered clinically significant by the investigator
16. Hemoglobin A1c (HgbA1c) greater than (>) 8 percent (%) (retesting is permitted if slightly elevated) or poorly controlled insulin-dependent diabetes (including hypoglycemic episodes). Participants may be rescreened after 3 months to allow optimization of diabetic control
17. Abnormally low serum vitamin B12 levels for the testing laboratory
18. History of human immunodeficiency virus (HIV) infection, history of hepatitis B infection within the past year, history of hepatitis C infection which has not been adequately treated, or history of spirochete infection of the central nervous system (example, syphilis, Lyme, or borreliosis)
19. Any other clinically significant abnormalities in physical examination, vital signs, laboratory tests, or ECG at Screening or Baseline which in the opinion of the investigator require further investigation or treatment or which may interfere with study procedures or safety
20. Malignant neoplasms within 3 years of Screening (except for basal or squamous cell carcinoma in situ of the skin, or localized prostate cancer in male participant, or localized breast cancer in female participants)
21. Answers "yes" to Columbia-Suicide Severity Rating Scale (C-SSRS) suicidal ideation Type 4 or 5, or any suicidal behavior assessment within 6 months before Screening, at Screening, or at the Baseline Visit, or has been hospitalized or treated for any suicidal behavior in lifetime
22. Known or suspected history of drug or alcohol abuse or dependence within 2 years before Screening or a positive urine drug test at Screening
23. Any other medical conditions (example, cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator could affect the participant's safety or interfere with the study assessments
24. Concurrent participation in a clinical study involving any anti-amyloid therapies (including any mAb therapies) within 6 months before Screening
25. Concurrent participation in a clinical study involving any anti-tau therapies
26. Participated in any other investigational medication or device study in the 3 months or 5 half-lives (whichever is longer) of the medication before Screening
27. Planned surgery which requires general anesthesia that would take place during the study
28. Visual or hearing impairment that would prevent the participant from performing psychometric tests accurately

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - UC San Diego Altman Clinical and Translational Research Insititute Clinic, La Jolla, California
  - Indiana University School of Medicine, Health Partners, Adult Neurology Clinic, Indianapolis, Indiana
- National Hospital for Neurology and Neurosurgery (NHNN) University College London(UCL) Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in the United States and United Kingdom from 28 June 2021 and 24 May 2024.
Pre-assignment Details: The study was conducted in two cohorts (Cohort A [Phase 1b and 2] and Cohort B). A total of 11 participants were screened, of which 3 were screen failures and 8 were enrolled to receive study treatment.
Groups:
- Cohort A: E2814: Participants received E2814 intravenous (IV) infusion, every 4 weeks (Q4W) at dose of 750 milligrams (mg) for 12 weeks, followed by 1500 mg for 12 weeks, further followed by 3000 mg for 12 weeks and then 4500 mg for up to 72 weeks.
- Cohort B: E2814: Participants received E2814 3000 mg, IV infusion, Q4W for 52 weeks.
Period: Overall Study
Arm/Group | Cohort A: E2814 | Cohort B: E2814
Started | 7 | 1
Cohort A: E2814 750 mg (Participants received E2814 750 mg, IV infusion, Q4W for 12 weeks in Phase 1b of Cohort A.) | 7 | 0
Cohort A: E2814 1500 mg (Participants received E2814 1500 mg, IV infusion, Q4W for 12 weeks in Phase 2 of Cohort A.) | 7 | 0
Cohort A: E2814 3000 mg (Participants received E2814 3000 mg, IV infusion, Q4W for 12 weeks in Phase 2 of Cohort A.) | 7 | 0
Cohort A: E2814 4500 mg (Participants received E2814 4500 mg, IV infusion, Q4W for 72 weeks in Phase 2 of Cohort A.) | 4 | 0
Completed | 2 | 0
Not Completed | 5 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Subject choice | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment.
Groups:
- Cohort A: E2814: Participants received E2814 IV infusion, Q4W at dose of 750 mg for 12 weeks, followed by 1500 mg for 12 weeks, further followed by 3000 mg for 12 weeks and then 4500 mg for up to 72 weeks.
- Total: Total of all reporting groups
Arm/Group | Cohort A: E2814 | Cohort B: E2814 | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 1 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: A TEAE was defined as adverse event (AE) that started at or after the time of administration of study drug or a worsening of severity from Baseline on or after 1st dose up to last assessment. An AE was any untoward medical occurrence in a participant or clinical investigation participant administered an investigational product. An AE did not necessarily have a causal relationship with the medicinal product. SAE was any untoward medical occurrence that at any dose: resulted in death; was life-threatening (that is, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Time Frame: From first dose of study drug up to 120 weeks
Population: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. As pre-specified in statistical analysis plan (SAP), the data of Cohort B was combined with Cohort A for E2814 3000 mg group due to same dosing in both cohorts.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: E2814 750 mg: Participants received E2814 750 mg, IV infusion, Q4W for 12 weeks.
- Cohort A: E2814 1500 mg: Participants received E2814 1500 mg, IV infusion, Q4W for 12 weeks.
- Cohort A+B: E2814 3000 mg: Participants received E2814 3000 mg, IV infusion, Q4W for 12 weeks in Cohort A and for 52 weeks in Cohort B.
- Cohort A: E2814 4500 mg: Participants received E2814 4500 mg, IV infusion, Q4W for up to 72 weeks.
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 8 | 4
Participants
  TEAEs | 4 | 1 | 8 | 4
  Serious TEAEs | 0 | 0 | 2 | 1

2. Primary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: Clinical laboratory tests included hematology, clinical chemistry, and urinalysis assessments. Markedly abnormal value was defined as a post-baseline value with an increase from baseline to a grade of 2 or higher on Common Terminology Criteria for Adverse events (CTCAE) Version 5.0 scale.
Time Frame: From first dose of study drug up to 120 weeks
Population: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. As pre-specified in SAP, the data of Cohort B was combined with Cohort A for E2814 3000 mg group due to same dosing in both cohorts.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 8 | 4
Participants | 0 | 1 | 1 | 2

3. Primary Outcome: Number of Participants With Clinically Significant Change in Vital Signs Values
Description: Vital sign measurements included systolic and diastolic blood pressure, pulse, respiratory rate, body temperature, height and weight assessment. The clinically significant assessment was based on investigator judgement.
Time Frame: From first dose of study drug up to 120 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 8 | 4
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings
Description: The clinically significant assessment was based on investigator judgement.
Time Frame: From first dose of study drug up to 120 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 8 | 4
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Cohort A: Change From Baseline in Cerebrospinal Fluid (CSF) Free, CSF Bound and Total Microtubule Binding Region of Tau (MTBR-tau; Starting at Amino Acid 354 and 299) at 12 Weeks
Description: Total MTBR-Tau was the total of bound MTBR-Tau + free MTBR-Tau. CSF samples were collected for the assessment.
Time Frame: Pre-dose at Week 12
Population: The Pharmacodynamic (PD) Analysis Set was the group of participants who received at least 1 dose of study drug and had sufficient PD data to derive at least 1 PD parameter. As planned, this outcome measure was assessed for E2814 750 mg only in Cohort A.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort A: E2814 750 mg
Number analyzed (Participants) | 7
nanogram per milliliter (ng/mL)
  Change in CSF Free MTBR-tau354 | -0.0534 (0.0690)
  Change in CSF Free MTBR-tau299 | -0.0147 (0.0267)
  Change in CSF Bound MTBR-tau354 | 0.178 (0.0886)
  Change in CSF Bound MTBR-tau299 | 0.0420 (0.0194)
  Change in CSF Total MTBR-tau354 | 0.125 (0.0899)
  Change in CSF Total MTBR-tau299 | 0.0273 (0.0191)

6. Secondary Outcome: Cohort A, Cmax: Maximum Observed Plasma Concentration for E2814
Description: The concentration of E2814 were measured by validated electrochemiluminescence assay methods and/or by a validated immunoprecipitation/purification followed by liquid chromatography with tandem mass spectrometry methods.
Time Frame: Cohort A, E2814 750 mg: Day 1 pre-dose up to 25 hours post-dose; Cohort A, E2814 1500 mg: Day 85 pre-dose up to 25 hours post-dose
Population: The Pharmacokinetic (PK) Analysis Set was the group of participants who received at least 1 dose of test drug and had sufficient PK data to derive at least 1 PK parameter. As planned, this PK parameter was assessed for E2814 750 mg and 1500 mg only in Cohort A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 7
microgram per milliliter (mcg/mL) | 218 (25.9) | 499 (24.3)

7. Secondary Outcome: Cohort A, Tmax: Time to Reach the Maximum Plasma Concentration for E2814
Description: The concentration of E2814 was measured by validated electrochemiluminescence assay methods and/or by a validated immunoprecipitation/purification followed by liquid chromatography with tandem mass spectrometry methods.
Time Frame: as for outcome 6
Population: The PK Analysis Set was the group of participants who received at least 1 dose of test drug and had sufficient PK data to derive at least 1 PK parameter. As planned, this PK parameter was assessed for E2814 750 mg and 1500 mg only in Cohort A.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 7
hours | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 5.00]

8. Secondary Outcome: Cohort A, AUC(0-672h): Area Under the Plasma Concentration-time Curve From Zero Time to 672 Hours for E2814
Description: as for outcome 7
Time Frame: Cohort A, E2814 750 mg: Day 1 pre-dose up to 672 hours post-dose; Cohort A, E2814 1500 mg: Day 85 pre-dose up to 672 hours post-dose
Population: PK Analysis Set was group of participants who received at least 1 dose of test drug and had sufficient PK data to derive at least 1 PK parameter. As planned, this PK parameter was assessed for E2814 750 mg and 1500 mg only in Cohort A. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure (sampling for first dose of 1500 mg was less intense versus the first dose of 750 mg; thus, no participants were evaluable for 1500 mg group for AUC[0-672h]).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 0
hour*microgram per milliliter (h*mcg/mL) | 66500 (23.2) |

9. Secondary Outcome: Cohort A, Cmax: Maximum Observed Serum Concentration for E2814
Description: as for outcome 7
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 7
mcg/mL | 41.7 (64.1) | 101 (47.1)

10. Secondary Outcome: Cohort A, Tmax: Time to Reach the Maximum Serum Concentration for E2814
Description: as for outcome 7
Time Frame: as for outcome 6
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 7
hours | 1.00 [1.00 to 25.00] | 5.00 [1.00 to 9.00]

11. Secondary Outcome: Cohort A, AUC(0-672h): Area Under the Serum Concentration-time Curve From Zero Time to 672 Hours for E2814
Description: as for outcome 7
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg
Number analyzed (Participants) | 7 | 0
h*mcg/mL | 8030 (54.8) |

12. Secondary Outcome: Cohort A: CSF Concentrations of E2814
Description: as for outcome 7
Time Frame: Pre-dose at Days 1, 84, 85, 169, 253, 421, and 757
Population: The PK Analysis Set was the group of participants who received at least 1 dose of test drug and had sufficient PK data to derive at least 1 PK parameter. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable at given time points for specified dosing group.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort A: E2814 3000 mg: Participants received E2814 3000 mg, IV infusion, Q4W for 12 weeks.
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 5 | 2
ng/mL
  Day 1: Pre-dose: number analyzed (Participants) | 7 | 0 | 0 | 0
  Day 1: Pre-dose | 0 (0) |  |  |
  Day 84: Pre-dose: number analyzed (Participants) | 2 | 0 | 0 | 0
  Day 84: Pre-dose | 172 (77.8) |  |  |
  Day 85: Pre-dose: number analyzed (Participants) | 5 | 0 | 0 | 0
  Day 85: Pre-dose | 153 (32.2) |  |  |
  Day 169: Pre-dose: number analyzed (Participants) | 0 | 7 | 0 | 0
  Day 169: Pre-dose |  | 429 (212) |  |
  Day 253: Pre-dose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Day 253: Pre-dose |  |  | 806 (426) |
  Day 421: Pre-dose: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 421: Pre-dose |  |  | 1035 (35.4) |
  Day 757: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Day 757: Pre-dose |  |  |  | 1611 (1567)

13. Secondary Outcome: Number of Participants With Treatment-emergent Positive Serum Anti-E2814 Antibody
Description: Anti-E2814 antibodies were measured by validated electrochemiluminescence assay.
Time Frame: From first dose of study drug up to 120 weeks
Population: The Safety Analysis Set was the group of participants who received at least 1 dose of study drug and had at least 1 post-dose safety assessment. As pre-specified in SAP, the data of Cohort B was combined with Cohort A for E2814 3000 mg group due to same dosing in both cohorts. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 6 | 3
Participants | 1 | 1 | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Positive Plasma Anti-E2814 Antibody
Description: Anti-E2814 antibodies were measured by validated electrochemiluminescence assay.
Time Frame: From first dose of study drug up to 120 weeks
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 7 | 7 | 6 | 3
Participants | 1 | 1 | 1 | 1

15. Secondary Outcome: Cohort A: Change From Baseline in CSF Concentrations of Total MTBR-tau243
Description: CSF samples were collected for the assessment.
Time Frame: Baseline, and pre-dose at Days 84, 169, 253, 421, 505, 589, and 757
Population: The PD Analysis Set was the group of participants who received at least 1 dose of study drug and had sufficient PD data to derive at least 1 PD parameter. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies participants evaluable at given time points for specified dosing group.
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 2 | 5 | 4 | 2
picogram per milliliter (pg/mL)
  Change at Day 84: Pre-dose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change at Day 84: Pre-dose | -210 (156) | -139 (53.5) |  |
  Change at Day 169: Pre-dose: number analyzed (Participants) | 0 | 1 | 3 | 0
  Change at Day 169: Pre-dose |  | -151 (NA) — Standard Deviation could not be calculated for single participant. | -236 (88.3) |
  Change at Day 253: Pre-dose: number analyzed (Participants) | 0 | 0 | 4 | 0
  Change at Day 253: Pre-dose |  |  | -296 (232) |
  Change at Day 421: Pre-dose: number analyzed (Participants) | 0 | 0 | 2 | 0
  Change at Day 421: Pre-dose |  |  | -216 (127) |
  Change at Day 505: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change at Day 505: Pre-dose |  |  |  | -315 (NA) — Standard Deviation could not be calculated for single participant.
  Change at Day 589: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change at Day 589: Pre-dose |  |  |  | -147 (NA) — Standard Deviation could not be calculated for single participant.
  Change at Day 757: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change at Day 757: Pre-dose |  |  |  | -381 (377)

16. Secondary Outcome: Cohort A: Change From Baseline in CSF Concentrations of Phosphorylated Tau (P-tau) 181, 205, and 217
Description: CSF samples were collected for the assessment.
Time Frame: Baseline, and pre-dose at Days 84, 169, 253, 421, 505, 589, and 757
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 2 | 5 | 5 | 2
pg/mL
  Change in P-tau 181 at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau 181 at Day 84: Predose | -166.50 (33.177) | 2.41 (204.061) |  |
  Change in P-tau 181 at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau 181 at Day 169: Predose |  | -10.32 (131.136) | -249.82 (351.972) |
  Change in P-tau 181 at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau 181 at Day 253: Predose |  |  | -308.74 (443.284) |
  Change in P-tau 181 at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau 181 at Day 421: Predose |  |  | -84.85 (106.021) | -1032.26 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 181 at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 181 at Day 505: Predose |  |  |  | -50.49 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 181 at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 181 at Day 589: Predose |  |  |  | -106.21 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 181 at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau 181 at Day 757: Predose |  |  |  | -606.64 (561.342)
  Change in P-tau 205 at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau 205 at Day 84: Predose | -38.37 (26.736) | -14.70 (101.226) |  |
  Change in P-tau 205 at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau 205 at Day 169: Predose |  | -67.43 (126.128) | -34.19 (86.949) |
  Change in P-tau 205 at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau 205 at Day 253: Predose |  |  | -84.42 (71.648) |
  Change in P-tau 205 at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau 205 at Day 421: Predose |  |  | -25.26 (4.975) | -113.91 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 205 at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 205 at Day 505: Predose |  |  |  | -24.12 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 205 at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 205 at Day 589: Predose |  |  |  | 4.48 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 205 at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau 205 at Day 757: Predose |  |  |  | -73.59 (58.215)
  Change in P-tau 217 at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau 217 at Day 84: Predose | -190.56 (120.537) | -216.52 (258.741) |  |
  Change in P-tau 217 at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau 217 at Day 169: Predose |  | -294.28 (350.271) | -188.49 (47.791) |
  Change in P-tau 217 at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau 217 at Day 253: Predose |  |  | -375.74 (246.487) |
  Change in P-tau 217 at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau 217 at Day 421: Predose |  |  | -217.44 (134.880) | -680.92 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 217 at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 217 at Day 505: Predose |  |  |  | -368.02 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 217 at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau 217 at Day 589: Predose |  |  |  | -135.13 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau 217 at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau 217 at Day 757: Predose |  |  |  | -422.60 (335.717)

17. Secondary Outcome: Cohort A: Change From Baseline in Ratio of CSF Concentrations of p-Tau/Non-phosphorylated (np) Tau for 181, 217, and 205
Description: CSF samples were collected for the assessment.
Time Frame: Baseline, and pre-dose at Days 84, 169, 253, 421, 505, 589, and 757
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A: E2814 3000 mg | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 2 | 5 | 5 | 2
ratio
  Change in P-tau181/np-tau181 ratio at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau181/np-tau181 ratio at Day 84: Predose | 0.95 (2.463) | 10.21 (12.187) |  |
  Change in P-tau181/np-tau181 ratio at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau181/np-tau181 ratio at Day 169: Predose |  | 17.54 (16.734) | -8.88 (15.713) |
  Change in P-tau181/np-tau181 ratio at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau181/np-tau181 ratio at Day 253: Predose |  |  | 2.96 (12.693) |
  Change in P-tau181/np-tau181 ratio at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau181/np-tau181 ratio at Day 421: Predose |  |  | 3.23 (4.146) | -8.78 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau181/np-tau181 ratio at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau181/np-tau181 ratio at Day 505: Predose |  |  |  | 11.64 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau181/np-tau181 ratio at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau181/np-tau181 ratio at Day 589: Predose |  |  |  | 0.40 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau181/np-tau181 ratio at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau181/np-tau181 ratio at Day 757: Predose |  |  |  | -6.87 (7.470)
  Change in P-tau205/np-tau205 ratio at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau205/np-tau205 ratio at Day 84: Predose | 0.42 (0.950) | 3.51 (2.221) |  |
  Change in P-tau205/np-tau205 ratio at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau205/np-tau205 ratio at Day 169: Predose |  | 2.08 (0.525) | 0.86 (4.695) |
  Change in P-tau205/np-tau205 ratio at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau205/np-tau205 ratio at Day 253: Predose |  |  | 2.53 (1.647) |
  Change in P-tau205/np-tau205 ratio at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau205/np-tau205 ratio at Day 421: Predose |  |  | 1.16 (0.915) | 4.53 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau205/np-tau205 ratio at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau205/np-tau205 ratio at Day 505: Predose |  |  |  | 2.32 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau205/np-tau205 ratio at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau205/np-tau205 ratio at Day 589: Predose |  |  |  | 2.02 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau205/np-tau205 ratio at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau205/np-tau205 ratio at Day 757: Predose |  |  |  | 1.80 (0.035)
  Change in P-tau217/np-tau217 ratio at Day 84: Predose: number analyzed (Participants) | 2 | 5 | 0 | 0
  Change in P-tau217/np-tau217 ratio at Day 84: Predose | -3.03 (4.624) | -5.49 (4.240) |  |
  Change in P-tau217/np-tau217 ratio at Day 169: Predose: number analyzed (Participants) | 0 | 3 | 3 | 0
  Change in P-tau217/np-tau217 ratio at Day 169: Predose |  | -8.13 (5.564) | -8.48 (6.258) |
  Change in P-tau217/np-tau217 ratio at Day 253: Predose: number analyzed (Participants) | 0 | 0 | 5 | 0
  Change in P-tau217/np-tau217 ratio at Day 253: Predose |  |  | -10.74 (5.265) |
  Change in P-tau217/np-tau217 ratio at Day 421: Predose: number analyzed (Participants) | 0 | 0 | 2 | 1
  Change in P-tau217/np-tau217 ratio at Day 421: Predose |  |  | -10.16 (4.143) | -15.35 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau217/np-tau217 ratio at Day 505: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau217/np-tau217 ratio at Day 505: Predose |  |  |  | -16.05 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau217/np-tau217 ratio at Day 589: Predose: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change in P-tau217/np-tau217 ratio at Day 589: Predose |  |  |  | -8.52 (NA) — Standard Deviation could not be calculated for single participant.
  Change in P-tau217/np-tau217 ratio at Day 757: Predose: number analyzed (Participants) | 0 | 0 | 0 | 2
  Change in P-tau217/np-tau217 ratio at Day 757: Predose |  |  |  | -14.56 (5.138)

18. Secondary Outcome: Cohort A: Change From Baseline in Tau Positron Emission Tomography (PET) Standardized Uptake Value Ratio (SUVR) by Region
Description: Tau-PET imaging uses radiotracers to visualize tau protein deposits in the brain for regional assessment of tau pathology. SUVR is ratio of tracer uptake in each of the cingulate, frontal, medial, occipital, parietal, whole cortical, meta temporal, and temporal cortices relative to tracer uptake in the cerebellum.
Time Frame: Baseline, at Weeks 60 and 108
Population: The PD Analysis Set was the group of participants who received at least 1 dose of study drug and had sufficient PD data to derive at least 1 PD parameter. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure. As planned, this outcome measure was assessed for 4500 mg only in Cohort A.
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Cohort A: E2814 4500 mg
Number analyzed (Participants) | 3
SUVR
  Change in PET tau SUVR in Cingulate Region at Week 60 | 0.135 (0.3756)
  Change in PET tau SUVR in Cingulate Region at Week 108 | 0.296 (0.4628)
  Change in PET tau SUVR in Frontal Region at Week 60 | 0.138 (1.0103)
  Change in PET tau SUVR in Frontal Region at Week 108 | 0.159 (0.9609)
  Change in PET tau SUVR in Medial Temporal Region at Week 60 | 0.165 (0.5615)
  Change in PET tau SUVR in Medial Temporal Region at Week 108 | 0.071 (0.5421)
  Change in PET tau SUVR in Occipital Region at Week 60 | 0.258 (0.9359)
  Change in PET tau SUVR in Occipital Region at Week 108 | 0.320 (0.8409)
  Change in PET tau SUVR in Parietal Region at Week 60 | 0.124 (0.9826)
  Change in PET tau SUVR in Parietal Region at Week 108 | 0.017 (0.8415)
  Change in PET tau SUVR in Temporal Region at Week 60 | 0.218 (0.9283)
  Change in PET tau SUVR in Temporal Region at Week 108 | 0.093 (0.7699)
  Change in PET tau SUVR in Meta-Temporal Region at Week 60 | 0.179 (0.9515)
  Change in PET tau SUVR in Meta-Temporal Region at Week 108 | 0.014 (0.7942)
  Change in PET tau SUVR in Whole Cortical Gray Matter (GM) Region at Week 60 | 0.172 (0.9461)
  Change in PET tau SUVR in Whole Cortical GM Region at Week 108 | 0.133 (0.8421)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 120 weeks
Description: As pre-specified in SAP, the data of Cohort B was combined with Cohort A for E2814 3000 mg group due to same dosing in both cohorts.
Arm/Group | Cohort A: E2814 750 mg | Cohort A: E2814 1500 mg | Cohort A+B: E2814 3000 mg | Cohort A: E2814 4500 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 2/8 | 1/4
Other Adverse Events (participants affected / at risk) | 4/7 | 1/7 | 7/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: E2814 750 mg (N=7) | Cohort A: E2814 1500 mg (N=7) | Cohort A+B: E2814 3000 mg (N=8) | Cohort A: E2814 4500 mg (N=4)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: E2814 750 mg (N=7) | Cohort A: E2814 1500 mg (N=7) | Cohort A+B: E2814 3000 mg (N=8) | Cohort A: E2814 4500 mg (N=4)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemiapraxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic pigmented purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT04971733/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT04971733/SAP_001.pdf